CLINICAL TRIAL: NCT05700331
Title: Fecal Microbiota Transplantation for Patients With Chronic Widespread Pain: A Pilot Prospective Single-arm Interventional Study
Brief Title: Fecal Microbiota Transplantation for Patients With Chronic Widespread Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending for funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Regina Wing Shan Sit, Prof. Regina Wing Shan SIT, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022.295
Record Dates: First submitted 2022-12-23; First posted 2023-01-26 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Chronic Widespread Pain
Keywords: Gut Microbiota; Fecal Microbiota Transplantation
MeSH Terms: conditions — Chronic Pain | interventions — Fecal Microbiota Transplantation; Sigmoidoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chronic Widespread Pain patients (Experimental): 3 FMT infusions, 2 weeks apart Procedures for Infusion: 100-200 ml of FMT solution or sterile saline will be infused over 2-3 minutes into the distal duodenum or jejunum via oesophago-gastro-duodenoscopy (OGD). After infusion, subjects will be monitored for 1 hour before discharged.
  Interventions: Procedure: Fecal Microbiota Transplantation; Procedure: Sigmoidoscopy

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — FMT performed at week 0, week-2 and week-4: FMT solution will be prepared using stool from a single donor or mixing of stool from multiple donors. Feces will be diluted with sterile saline (0.9%). This solution will be blended and strained with filter. The resulting supernatant will then be used directly as fresh FMT solution or stored as frozen FMT solution for future FMT.
  Procedures for Infusion: 100-200 ml of FMT solution or sterile saline will be infused over 2-3 minutes into the distal duodenum or jejunum via oesophago-gastro-duodenoscopy (OGD). After infusion, subjects will be monitored for 1 hour before discharged.
  2 study biopsies in total (from duodenum) will be obtained during FMT infusion via OGD.
Procedure: Sigmoidoscopy — Optional sigmoidoscopy will be done at week 0 and week 4, during which 2 study biopsies in total (obtained via sigmoidoscopy) will be obtained from the rectum.

SUMMARY:
This study aims to explore the effect of Fecal Microbiota Transplantation (FMT) on the clinical symptomatology in Chronic Widespread Pain (CWP), to assess the acceptability, tolerability, and safety of FMT in patients with CWP, as well as explore the effect of FMT on the gut microbiome diversity in CWP. The investigators hypothesize that fecal microbiota transplantation will reduce pain intensity in patients with CWP, is acceptable, safe, and tolerable in patients with CWP, and will achieve change of gut microbiome diversity after FMT treatment.

DETAILED DESCRIPTION:
In this proposed proof-of-concept pilot study, the investigators capitalize an establish chronic pain cohort to explore the effect of FMT in improving the pain symptomology in patients with CWP. This will be a 12-week single-arm prospective interventional study, all study subjects will receive 3 FMT infusions (N =20).

ELIGIBILITY:
Inclusion Criteria:

• Participants aged ≥ 18 with diagnosis CWP; A modified version of the London Fibromyalgia Epidemiology Study Screening Questionnaire (LFESSQ) will be used to screen for the presence of CWP.

Exclusion Criteria:

* Patients with fibromyalgia, a subgroup with complex neurobiological, behavioural and psychological factors on its pathogenesis, will be excluded.[8] This will be based on The American College of Rheumatology 2010 when subjects with CWP but with a widespread pain index (WPI) of ≥ 7 and a symptom severity scale (SSS) score of ≥ 5 or a WPI between 3 and 6 and an SSS score of ≥ 9.
* Patients have a history of inflammatory bowel disease or gastrointestinal malignancy
* Patients have previous abdominal surgery (other than cholecystectomy or appendectomy)
* Patients have depression defined by having a Patient Health Questionnaire-9 (PHQ-9) score > 15
* Patients have anxiety defined by having a Generalized Anxiety Disorder 7 (GAD7) score > 10
* Patients have active infection at the time of inclusion
* Patients have used antibiotic therapy or anti-inflammatory drugs within the past 7 days
* Patients have any other organic causes that can explain the symptoms of CWP
* Current pregnancy
* Confirmed current active malignancy or cancers
* Pregnancy test negative for all female patients of child-bearing potential (except postmenopausal patients and sterilized patients).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Changes in self-reported pain severity | Study week 0 , 6 , 12
  Pain severity will be measured by Brief Pain Inventory (BPI), which consists of 4-item severity and 7-item interference subscale scores (Score range 0-10)

SECONDARY OUTCOMES:
Safety and tolerability of supplementation of FMT | through study completion, an average of 1 year
  Adverse events will be monitored throughout the study
Changes in objectively measured pain pressure threshold | Study week 0 , 6 , 12
  Fischer pressure algometer will be used for measuring pain pressure threshold (PPT).
Changes in comorbid psychopathology (anxiety symptoms) | Study week 0 , 6 , 12
  The Generalized Anxiety Disorder (GAD-7, score range 0-21) will be used to measure anxiety status
Changes in comorbid psychopathology (depressive symptoms) | Study week 0 , 6 , 12
  The Patient Health Questionnaire (PHQ-9, score range 0-27) will be used to measure anxiety status
Changes in health-related quality of life | Study week 0 , 6 , 12
  The overall the health-related quality of life (HRQoL) will be measured by the EuroQoul-5 dimensions questionnaire (EQ-5D-5L)
Changes in Alpha diversity index of gut microbiota | Study week 0 , 6 , 12
  Alpha diversity of the gut microbiome using the Shannon's and inverse Simpson indices will be computed from the operational taxonomic units (OTUs)
Sociodemographic data | At baseline, Study week 0
  Demographics and medical history such as sex, age, smoking and alcohol status, disease onset, co-morbid illness, drug history, clinical test results will be obtained by reviewing of patient medical notes and interview with patients by doctors and research staff

OTHER OUTCOMES:
Blood sample (Full blood count) | Study week 0, 2, 4, 6, 12
  Not more than 20ml of blood will be collected
Number of participants with With Laboratory Values (Biochemistry profile) | Study week 0, 2, 4, 6, 12
  Not more than 20ml of blood will be collected
Blood sample (C-reactive protein) | Study week 0, 2, 4, 6, 12
  Not more than 20ml of blood will be collected
Stool sample | Study week 0, 6, 12
  Stool sample collected through stool sample collection kit with Norgen preservation solutions

CONTACTS AND LOCATIONS:
Overall Officials: Regina Wing Shan Sit, MD, Principal Investigator — The Jockey Club School of Public Health and Primary Care, Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Shatin, Hong Kong